CLINICAL TRIAL: NCT06314763
Title: Rivaroxaban Sotorasib Interaction Study
Acronym: ROSIE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ROSIE
Record Dates: First submitted 2024-02-05; First posted 2024-03-18 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-01

CONDITIONS: Drug Drug Interaction Study
Keywords: Lung cancer; Non small cell lung cancer; NSCLC; Sotorasib; Lumykras; Lumakras; Rivaroxaban; Xarelto; DOAC; Enzyme inhibitors; Molecular Mechanisms of Pharmacological Action; Venous thromboembolism
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Venous Thromboembolism | interventions — Rivaroxaban; sotorasib

STUDY DESIGN:
Intervention Model Description: An open label single-sequence pharmacokinetic drug-drug interaction study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Single dose rivaroxaban 20 mg and steady-state sotorasib 960 mg (Experimental): To assess the pharmacokinetics of single dose rivaroxaban in presence and absence of 960 mg sotorasib at pharmacokinetic steady-state. Samples will be taken pre-dose (t=0) and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, and 48 hours post ingestion.
  Interventions: Drug: Rivaroxaban 20mg; Drug: Sotorasib 960mg

INTERVENTIONS:
Drug: Rivaroxaban 20mg — Single dose on day 1 and day 16
  Other Names: Xarelto
Drug: Sotorasib 960mg — Daily dose from day 3 till day 16
  Other Names: Lumykras

SUMMARY:
Venous thromboembolic Events (VTEs) are common in lung cancer patients with an incidence of >15%, requiring anticoagulant treatment or prophylaxis. Although direct acting oral anticoagulants (DOACs) are the agents of first choice due to ease and patient friendliness, these drugs are often avoided in cancer patients due to suspected pharmacokinetic drug-drug interactions with oncolytic drugs. Sotorasib is the first KRASG12C inhibitor that has been approved by the US [FDA] and EU [EMA] for the treatment of adult patients with KRAS G12C-mutated locally advanced or metastatic NSCLC. Sotorasib has a potential to cause CYP3A-mediated drug-drug interactions due to induction of CYP3A and inhibition of P-GP. Rivaroxaban is the most frequently prescribed DOAC in the Netherlands. As rivaroxaban is a substrate for this enzyme and efflux pump, sotorasib may increase or decrease the exposure to rivaroxaban and, thus, impact its benefit-to-risk ratio. To enable safe combination of sotorasib and rivaroxaban, it is pivotal to investigate the magnitude of the pharmacokinetic interaction between these drugs.

DETAILED DESCRIPTION:
Objective:

To assess the pharmacokinetics of single dose rivaroxaban in presence and absence of 960 mg sotorasib at pharmacokinetic steady-state

Main study parameters/endpoints:

The geometric mean ratios of area under the concentration time curve (AUC) and maximum concentration (Cmax) of rivaroxaban in absence and presence of sotorasib, and their corresponding 90% confidence intervals.

Study design:

An open label single-sequence pharmacokinetic drug-drug interaction study in healthy volunteers.

Study population:

Healthy human volunteers aged between 18 and 65. Volunteers can't participate in this study if they have an increased risk for bleeding or blood clotting. Furthermore, volunteers receiving concomitant drugs with a pharmacokinetic or pharmacodynamic interaction with the investigational medicinal products will also be excluded.

Intervention:

The pharmacokinetics of a single dose rivaroxaban are assessed in presence and absence of sotorasib. The study participants will receive rivaroxaban (20 mg single dose ingested with food) on day 1, followed by a wash-out period on day 1 and 2, followed by daily administration of sotorasib 960 mg once daily on day 3-16 and rivaroxaban (20 mg single dose ingested with food) on day 16.

The pharmacokinetics of rivaroxaban will be assessed at T=0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 and 48 hours after administration on the days that rivaroxaban is administered.

The pharmacokinetics of sotorasib will be assessed at T=0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24h after administration on day 16.

Ethical consideration to the clinical trial including the expected benefit to the individual subject or group of patients represented by the study participants as well as the nature and extent of burden and risks: A drug-drug interaction study in patients on sotorasib is not considered feasible and methodologically sound, due to high co-morbidity and polypharmacy in patients with an indication for treatment with sotorasib. Single dose pharmacokinetic rivaroxaban studies in healthy volunteers are common and the gold standard to assess the impact of drug-drug interactions with DOACs. Single and multiple dose studies of sotorasib in healthy volunteers are considered and proven safe, likely due to high selectivity of the drug for KRAS G12C mutation that is only present in tumor cells of individuals with KRAS G12C mutated cancer. There is no individual benefit for participation in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 and not older than 65 years at screening.
2. Subject does not smoke more than 10 (e-)cigarettes, 2 cigars, or 2 pipes per day for at least 3 months prior to the first study day.
3. Subject has a Body Mass Index of 18 to 30 kg/m2 .
4. Subject is able and willing to sign the Informed Consent Form prior to screening evaluations.
5. Subject is in good age-appropriate health condition as established by medical history and physical examination within 4 weeks prior to day 1.
6. Subject has a normal blood pressure and pulse rate, according to the Investigator's judgement.

Exclusion Criteria:

1. An estimated glomerular filtration or creatinine clearance of less than 70mL/min.
2. Liver enzyme tests (ALAT, ASAT, GGT, total bilirubin, ALP) greater than 2 times the upper limit of normal.
3. Serum electrolytes (sodium, potassium, calcium, magnesium) outside the normal range of the NVKC reference ranges.
4. Hemocytometric values (hemoglobin, hematocrit, leukocytes, erythrocytes and thrombocytes) outside of the NVKC reference ranges.
5. A prothrombin time (PT) > 13.3 seconds.
6. An activated partial thromboplastin time (APTT) >38 seconds.
7. Clinically significant pathologies of the cardiovascular, bronchopulmonary, neuroendocrine systems, as well as diseases of the gastrointestinal tract, liver, kidneys and blood.
8. Documented history of sensitivity/idiosyncrasy to medicinal products or excipients.
9. Female subject is pregnant or lactating/breastfeeding or planning to become pregnant or breastfeed during treatment and for an additional 7 days after the last dose of sotorasib.
10. Female subjects of childbearing potential unwilling to use an effective method of contraception during treatment and for an additional 7 days after the last dose of sotorasib.
11. Male subjects with a female partner of childbearing potential who are unwilling to practice sexual abstinence (refrain from heterosexual intercourse) or use contraception during treatment and for an additional 7 days after the last dose of sotorasib.
12. Male subjects unwilling to abstain from donating sperm during treatment and for an additional 7 days after the last dose of sotorasib.
13. Consumption of foods and beverages containing poppy seeds, St. Johns Wort, grapefruit, or Seville oranges within 7 days prior to check-in.
14. Concomitant use of drugs, including herbs and food additives, with a pharmacokinetic or pharmacodynamic interaction, as assessed with most recent KNMP kennisbank and uptodate.com drug interaction databases.
15. Donation of plasma or blood (450ml or more) less than 2 months before start of the study.
16. Relevant history or current condition that might interfere with drug absorption, distribution, metabolism or excretion.
17. History of or current abuse of drugs or alcohol.
18. Inability to understand the nature and extent of the study and the procedures required.
19. Febrile illness within 3 days before Day 1.
20. History of internal bleeding of any genesis.
21. Known present congenital or acquired bleeding disorders.
22. History of liver disease.
23. History suggestive of esophageal (including esophageal spasm, esophagitis), gastric, or duodenal ulceration or bowel disease (including but not limited to peptic ulceration, gastrointestinal bleeding, ulcerative colitis, Crohn's disease, or irritable bowel syndrome); or a history of gastrointestinal surgery other than uncomplicated appendectomy.
24. Known gastrointestinal disease without active ulceration that can potentially lead to bleeding complications.
25. History of vascular retinopathy.
26. Known bronchiectasis.
27. History of pulmonary bleeding.
28. The following conditions known in medical history: coronary heart disease, previous cerebrovascular accident (CVA) or transient ischaemic attack.
29. Positive Hepatitis B Surface Antigen (HepBsAg) (indicative of chronic Hepatitis B or recent acute hepatitis B). Negative HepBsAg with a positive for hepatitis B core antibody (Hepatitis B core antibody testing is not required for screening, however if this is done and is positive, then hepatitis B surface antibody [anti-HBs] testing is necessary. Undetectable anti-HBs in this setting would suggest unclear and possible infection and needs exclusion).
30. Positive Hepatitis C virus antibody: Hepatitis C virus RNA by polymerase chain reaction (PCR) is necessary. Detectable Hepatitis C virus RNA suggests chronic hepatitis C.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-11-09 (Actual); Primary Completion 2024-03-21 (Actual); Study Completion 2024-03-21 (Actual)

PRIMARY OUTCOMES:
The pharmacokinetics (AUC) of single dose rivaroxaban in presence and absence of 960 mg sotorasib at pharmacokinetic steady-state. | 18 days
  The geometric mean ratios of area under the concentration time curve (AUC) of rivaroxaban in absence and presence of sotorasib, and their corresponding 90% confidence intervals. The pharmacokinetics of rivaroxaban will be assessed with standard compartmental or non-compartmental pharmacokinetic methods.
The pharmacokinetics (Cmax) of single dose rivaroxaban in presence and absence of 960 mg sotorasib at pharmacokinetic steady-state. | 18 days
  Maximum concentration (Cmax) of rivaroxaban in absence and presence of sotorasib, and their corresponding 90% confidence intervals. The pharmacokinetics of rivaroxaban will be assessed with standard compartmental or non-compartmental pharmacokinetic methods.

SECONDARY OUTCOMES:
The pharmacokinetics (AUC) of sotorasib in healthy volunteers. | 18 days
  Description of the area under the concentration time curve (AUC) of sotorasib at steady-state conditions in healthy volunteers, by means of standard compartmental or non-compartmental pharmacokinetic methods.
The pharmacokinetics (Cmax) of sotorasib in healthy volunteers. | 18 days
  Description of the maximum concentration (Cmax) of sotorasib at steady-state in healthy volunteers, by means of standard compartmental or non-compartmental pharmacokinetic methods.
Number of participants with treatment-related adverse events as assessed by CTCAE v6.0 | 18 days
  Description of the treatment-related events of sotorasib and rivaroxaban, graded with the most recent version (v6) of the Common Toxicity Criteria for Adverse Events (CTCAE)
Pharmacokinetic variability in AUC of rivaroxaban. | 18 days
  Assess the pharmacokinetic variability in area under the concentration time curve (AUC) of rivaroxaban between healthy subjects
Pharmacokinetic variability in Cmax of rivaroxaban. | 18 days
  Assess the pharmacokinetic variability in maximal concentration (Cmax) of rivaroxaban between healthy subjects
Pharmacokinetic variability in AUC of sotorasib. | 18 days
  Assess the pharmacokinetic variability in area under the concentration time curve (AUC) of sotorasib between healthy subjects.
Pharmacokinetic variability in Cmax of sotorasib. | 18 days
  Assess the pharmacokinetic variability in maximal concentration (Cmax) of sotorasib between healthy subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Rob ter Heine, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud university medical centre, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No